CLINICAL TRIAL: NCT03271151
Title: Effect of Duloxetine on Opioid Use After Total Knee Arthroplasty: A Double-blinded Randomized Control Trial
Brief Title: Effect of Duloxetine on Opioid Use After Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-0655
Record Dates: First submitted 2017-08-29; First posted 2017-09-01 (Actual); Results first posted 2022-04-26 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-09

CONDITIONS: Joint Disease; Pain, Acute; Pain, Chronic
MeSH Terms: conditions — Joint Diseases; Acute Pain; Chronic Pain | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Duloxetine ("Cymbalta") (Experimental): Epidural analgesia after knee arthroplasty is not as prevalent at HSS as formerly, in large part due to the rise of local infiltration analgesia. Studies using epidural analgesia may also lack generalizability given the infrequent use of epidural analgesia at other institutions. For these reasons, we plan to use adductor canal nerve blockade + local infiltration analgesia for management of immediate postoperative pain. Patients will receive spinal anesthesia as the primary anesthetic. It is particularly important to study duloxetine ("Cymbalta") in the context of local infiltration analgesia, as patients receiving local infiltration analgesia receive increased doses of opioids, compared to patients receiving epidural analgesia.
  Interventions: Drug: Cymbalta
- Placebo (Placebo Comparator): Placebo to compare pain scores and opioid use againts Duloxetine
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cymbalta — Duloxetine ("Cymbalta") is a serotonin and norepinephrine dual reuptake inhibitor (SNRI) that is an effective treatment for painful diabetic neuropathy. It is approved for major depressive disorder, generalized anxiety disorder, diabetic peripheral neuropathy, fibromyalgia, and chronic musculoskeletal pain
  Arms: Duloxetine ("Cymbalta")
Other: Placebo — Placebo to compare outcomes against Duloxetine
  Arms: Placebo

SUMMARY:
Post-discharge pain after total knee arthroplasty remains problematic; many patients have excessive pain at the 2 week time point (and often thereafter). Reduction in opioid use has become a national goal, due to the 'epidemic' in opioid misuse.

In addition to enrolling non-opioid users, we will enroll up to 15 chronic opioid users.

ELIGIBILITY:
Inclusion Criteria:

* Age 25 to 75 years
* Planned use of regional anesthesia
* Ability to follow study protocol
* English speaking (Primary outcome obtained via telephone call and secondary outcomes include questionnaires validated in English only)
* Patients planning on being discharged home or to a rehabilitation center that has agreed to participate

Exclusion Criteria:

* Current Use of duloxetine or other SNRIs, SSRIs, MAOIs, Tricyclic antidepressants, triptans (sumatriptan, rizatriptan, naratriptan, eletriptan, almotriptan, frovatriptan), lithium, buspirone, St. John's Wort
* Hepatic insufficiency

  o Hepatoxicity is reported as a side effect of duloxetine. "Median time to detection of transaminase elevation was about two months" (package insert 5.2
* Renal insufficiency (ESRD, HD, estimated creatinine clearance < 50 ml/min)

  * Severe CRI may impair duloxetine clearance
  * CLcr=[(140-age (years)] x weight (kg)x0.85 (for female patients)/[72xserum creatinine (mg/dL)]
* Patients younger than 25 years old and older than 75
* Patients intending to receive general anesthesia
* Allergy or intolerance to one of the study medications
* Patients with an ASA of IV
* Chronic gabapentin/pregabalin use (regular use for longer than 3 months)
* Patients with major prior ipsilateral open knee surgery.
* Chronic opioid use (taking opioids for longer than 3 months)

  * However, patients using chronic opioids may enroll in a parallel pilot study entitled 'effect of duloxetine on opioid use after total knee athroplasty among patients exposed to opioids- a pilot study'. The chronic opioid users will be allowed to continue their customary analgesics. The pilot study is otherwise identical to the main study.
  * This study will enroll up to 15 chronic opioid users. After that, all chronic opioid users are excluded.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2021-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques T YaDeau, MD, Phd, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Duloxetine ("Cymbalta") | Placebo
Started | 80 | 80
Completed | 78 | 77
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 1 | 3
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duloxetine ("Cymbalta") | Placebo | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 42 | 83
  >=65 years | 39 | 38 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (11) | 64 (7) | 63 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 35 | 75
  Male | 40 | 45 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 76 | 78 | 154
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Opioid Use
Description: Opioid use (measured in cumulative morphine equivalents)
Time Frame: Post-operative day 14
Measure: Mean (Standard Deviation); unit: Oral Morphine Equivalent (mg)
Arm/Group | Duloxetine ("Cymbalta") | Placebo
Number analyzed (Participants) | 78 | 77
Oral Morphine Equivalent (mg) | 288 (226) | 432.5 (374)

2. Primary Outcome: Pain Scores
Description: Numerical Rating Score pain with movement. Minimum value of 0, maximum value of 10. Higher scores mean more pain and worse outcome.
Time Frame: Post-operative day 14
Measure: Mean (Standard Deviation); unit: score on a scale (NRS)
Arm/Group | Duloxetine ("Cymbalta") | Placebo
Number analyzed (Participants) | 78 | 77
score on a scale (NRS) | 4.2 (2) | 4.8 (2.2)

3. Secondary Outcome: Pain Phenotype
Description: 2011 Survey Criteria for Fibromyalgia. Minimum value of 0, and maximum value of 12. A higher score means a worse outcome.
Time Frame: Day of surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Duloxetine ("Cymbalta") | Placebo
Number analyzed (Participants) | 80 | 80
score on a scale | 2 [1 to 4] | 2 [1 to 4]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Duloxetine ("Cymbalta") | Placebo
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80
Other Adverse Events (participants affected / at risk) | 2/80 | 3/80
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine ("Cymbalta") (N=80) | Placebo (N=80)
Hallucinations (General disorders) | 1 (1) | 1 (1) — Patient reported experiencing hallucinations. Unclear if related to study medication and/or opioid
Unable to Ejaculate (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Unclear if related to study medication and/or opioid medication
Increased diaphoresis, blood pressure, complaints of diarrhea decreased unration and tooth pain (General disorders) | 0 (0) | 1 (1) — Not typical duloxetine side effects; unclear if study related
Acne (General disorders) | 0 (0) | 1 (1) — Patient reported acne on chest and back, 14 days after surgery. Unclear if due to study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-27): https://cdn.clinicaltrials.gov/large-docs/51/NCT03271151/Prot_SAP_000.pdf